CLINICAL TRIAL: NCT05661578
Title: A Phase II, Single-Arm, Open-Label Study Evaluating the Safety and Pharmacokinetics of the Intravenous Fixed-Dose Combination (IV FDC) of Tiragolumab and Atezolizumab in Participants With Locally Advanced, Recurrent or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of the Intravenous Fixed-Dose Combination (IV FDC) of Tiragolumab and Atezolizumab in Participants With Locally Advanced, Recurrent or Metastatic Solid Tumors
Acronym: SKYSCRAPER-11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO44096; 2022-001157-23 (EudraCT Number); 2023-508489-14-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PD-L1-selected Solid Tumors
MeSH Terms: interventions — Tiragolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tiragolumab and Atezolizumab IV FDC (Experimental): Participants will receive tiragolumab and atezolizumab as an intravenous fixed dose combination (IV FDC) on Day 1 of each 21-day cycle until disease progression, loss of clinical benefit or unacceptable toxicity.
  Interventions: Drug: Tiragolumab and Atezolizumab IV FDC

INTERVENTIONS:
Drug: Tiragolumab and Atezolizumab IV FDC — Intravenous fixed dose combination (IV FDC) of tiragolumab 600 mg and atezolizumab 1200 mg once every 3 weeks (Q3W).

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics, and immunogenicity of tiragolumab and atezolizumab intravenous fixed-dose combination (IV FDC) in participants with histologically confirmed PD-L1-selected solid tumors whose disease is locally advanced, recurrent, or metastatic and for whom an investigational agent in combination with an anti-PD-L1 antibody is considered an acceptable treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy >=12 weeks
* Adequate hematologic and end organ function
* Recovery (i.e., improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia
* For female participants of childbearing potential, negative serum pregnancy test within 14 days prior to initiation of study treatment (Day 1 of Cycle 1)
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agree to refrain from donating eggs during the treatment period and for 5 months after the final dose of tiragolumab and atezolizumab IV FDC
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm during the treatment period and for 90 days after the final dose of tiragolumab and atezolizumab IV FDC to avoid exposing the embryo

Cancer-Specific Inclusion Criteria:

* Histologic documentation of locally advanced, recurrent, or metastatic malignancy, ineligible for definitive local therapy, for which a clinical trial of an investigational agent in combination with an anti-PD-L1 antibody is considered an acceptable treatment option. Participant must be informed of all standard of care options available for his/her cancer.
* No prior treatment with checkpoint inhibitor therapies (CPI-Naive)
* Measurable disease per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Submittal of archival tumor and/or fresh tumor tissue to the central laboratory for programmed death-1 (PD-L1) evaluation prior to enrollment
* PD-L1 selected tumors, as determined by the investigational VENTANA PD-L1 (SP263) immunohistochemistry (IHC) assay

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 5 months after the final dose of tiragolumab and atezolizumab IV FDC
* Significant cardiovascular disease
* Known clinically significant liver disease
* Poorly controlled Type 2 diabetes mellitus
* Major surgical procedure within 28 days prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure during the study
* Any other diseases, metabolic dysfunction, physical examination finding, and/or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or may render the participant at high risk from treatment complications
* History of autoimmune disease
* Treatment with systemic immunosuppressive medications within 2 weeks prior to Day 1 of Cycle 1
* History of idiopathic pulmonary fibrosis, pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Severe infections within 4 weeks prior to Day 1 of Cycle 1 or recent infections/oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1

Cancer-Specific Exclusion Criteria:

* Any anti-cancer therapy, whether investigational or approved within 3 weeks prior to initiation of study treatment
* Prior treatment with immune checkpoint inhibitors (CPIs)
* Less than 5 drug-elimination half-lives (~100 days for typical monoclonal antibody [Mab]) from the last dose of monoclonal antibodies (MAbs), and MAb-Derived Therapies (excluding CPIs) and the proposed Day 1 of Cycle 1
* Less than 6 weeks between the last dose of prior immunomodulators and the proposed Day 1 of Cycle 1
* Less than 6 weeks or 5-drug-elimination half-lives, whichever is shorter, of prior treatment with cancer vaccines and/or cytokines have elapsed between the last dose and the proposed Cycle 1, Day 1
* Any history of an immune-mediated Grade 4 adverse event attributed to prior cancer immunotherapy
* Any history of an immune-mediated Grade 3 adverse event attributed to prior cancer immunotherapy that resulted in permanent discontinuation of the prior immunotherapeutic agent and/or occurred </=6 months prior to Day 1 of Cycle 1
* Any immune-mediated adverse events related to prior cancer immunotherapy must have resolved completely to baseline
* Adverse events from prior anti-cancer therapy that have not resolved to Grade <=1 except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 24 months

SECONDARY OUTCOMES:
Area Under the Concentration Time Curve (AUC) of Tiragolumab | Cycle 1 (each cycle is 21 days): Days 1, 2, 8 and 15
AUC of Atezolizumab | Cycle 1 (each cycle is 21 days): Days 1, 2, 8 and 15
Maximum Serum Concentration (Cmax) of Tiragolumab | Cycle 1 (each cycle is 21 days): Days 1, 2, 8 and 15
Cmax of Atezolizumab | Cycle 1 (each cycle is 21 days): Days 1, 2, 8 and 15
Percentage of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab | Day 1 of Cycles (each cycle is 21 days) 1, 2, 3, 4, 8, 12, 16 and treatment discontinuation (TD) visit (up to approximately 24 months)
Percentage of Participants With ADAs to Atezolizumab | Day 1 of Cycles (each cycle is 21 days) 1, 2, 3, 4, 8, 12, 16 and TD visit (up to approximately 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- Medical Oncology Associates, Spokane, Washington, United States
- Chongqing Sanxia Central Hospital, Chongqing, China
- Croatia (2):
  - General Hospital Pula, Pula
  - Klinicki bolnicki centar Zagreb, Zagreb
- Greece (3):
  - IASO Obstetrics Gynecology Clinic, Marousi
  - University General Hospital of Patras, Pátrai
  - St. Luke's Hospital, Thessaloniki
- Serbia (3):
  - Oncomed-System, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
- Spain (9):
  - ICO l?Hospitalet ? Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Instituto de Investigacion Oncologica Vall dHebron (VHIO) - EPON, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - START MADRID_Hospital Universiario Fundacion Jimenez Diaz, Madrid
  - START Madrid_Hospital Universitario HM Sanchinarro_CIOCC, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - TAIPEI VETERANS GENERAL HOSPITAL, Urology, Taipei
- Turkey (Türkiye) (7):
  - Namik Kemal University, Alt?nova
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi University Medical Faculty, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Memorial Sisli Private Hospital, Istanbul
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
  - Medical Park Seyhan Hospital, Seyhan

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing